CLINICAL TRIAL: NCT01750034
Title: Best Method of Burn Wound Care: A Prospective Randomized Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility issues
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-2288
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Burns
Keywords: Burns; Wounds and injuries; Bandages
MeSH Terms: conditions — Burns; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Closed method (Active Comparator): Burn patients randomized to closed method of burn wound care.
  Interventions: Procedure: Closed method
- Open method (Experimental): Burn patients randomized to the open method of burn wound care.
  Interventions: Procedure: Open method

INTERVENTIONS:
Procedure: Closed method — Subjects will have their wounds managed by covering with gauze and changing this gauze 3 to 7 times per week.
  Other Names: Bandage method; Dressing method
  Arms: Closed method
Procedure: Open method — Subjects will have their burns managed by keeping the wounds exposed to the air.
  Other Names: Exposure method
  Arms: Open method

SUMMARY:
The purpose of this study is to better understand how to best care for burn wounds.

DETAILED DESCRIPTION:
Participants: Patients presenting to Kamuzu Central Hospital in Lilongwe Malawi with burn wounds occuring within 72 hours of admission.

Procedures (methods): This is a prospective randomized trial. Subjects will be randomized during admission to receive either open dressing care or closed dressing care of their burn wounds.

ELIGIBILITY:
Inclusion Criteria:

* Burn wound admitted to the hospital
* Signed informed consent
* Burn wound occuring within 72 hours of admission

Exclusion Criteria:

* Language other than Chichewa or English
* Inability to access of phone (required for follow-up)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Time to healing | 30-day
  Time from burn injury to healing (defined as at least 90% epithelialization) as determined by hospital records, outpatient clinical records and telephone contact (with subject or next-of-kin) per study protocol.

SECONDARY OUTCOMES:
Mortality | 30-day
  Mortality within 30 days of burn injury, as determined by hospital records, outpatient clinical records and telephone contact (with next-of-kin) per study protocol.
Burn wound infection rate | 30-day
  Clinical suspicion of infection defined by presence of (a) burn wound cellulitis (erythema and/or edema AND pain and/or tenderness at the border of the wound), or (b) burn wound infection (change in appearance of the burn including focal or multifocal brown, black or violaceous discoloration OR rapid separation of the eschar OR conversion of partial thickness to full thickness burn).

OTHER OUTCOMES:
Microbiologic profile of clinical infections | 30-day
  Qualitative microbiologic culture results and sensitivity panels from surface swabs taken from infected burn wounds (as defined by clinical criteria described in the secondary outcome "burn wound infection rate").
Number of surgical procedures | 30-day
  Number of surgical procedures required including indication and type of procedure.
percent skin graft survival | 30-day
  Percent survival (defined as area surviving / total area grafted at 7 days) of skin grafts.
Hospital length of stay | 30-day
  Length of stay during initial hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Jared Gallaher, MD, Principal Investigator — UNC Chapel Hill Department of Surgery

REFERENCES:
- [Background] Gosselin RA, Kuppers B. Open versus closed management of burn wounds in a low-income developing country. Burns. 2008 Aug;34(5):644-7. doi: 10.1016/j.burns.2007.09.013. Epub 2008 Jan 15. PMID 18226462
- [Background] Dominguez O, Bains JW, Lynch JB, Lewis SR. Treatment of burns with silver nitrate versus exposure method: analysis of 200 patients. Plast Reconstr Surg. 1967 Nov;40(5):489-93. doi: 10.1097/00006534-196711000-00012. No abstract available. PMID 6074149
- [Background] HOLMAN SP, SHAYA ES, HOFFMEISTER FS, EDGERTON MT Jr. Studies on burns. I. The exposure method vs. occlusive dressings in the local treatment of experimental burns. Ann Surg. 1956 Jan;143(1):49-56. doi: 10.1097/00000658-195601000-00006. No abstract available. PMID 13275898
- [Background] Kiser MM, Samuel JC, Mclean SE, Muyco AP, Cairns BA, Charles AG. Epidemiology of pediatric injury in Malawi: burden of disease and implications for prevention. Int J Surg. 2012;10(10):611-7. doi: 10.1016/j.ijsu.2012.10.004. Epub 2012 Nov 7. PMID 23142508
- [Background] Samuel JC, Campbell EL, Mjuweni S, Muyco AP, Cairns BA, Charles AG. The epidemiology, management, outcomes and areas for improvement of burn care in central Malawi: an observational study. J Int Med Res. 2011;39(3):873-9. doi: 10.1177/147323001103900321. PMID 21819720